CLINICAL TRIAL: NCT06407609
Title: Positive Outcomes of the Supplementation With Lecithin-based Delivery Form of Curcuma Longa and of Boswellia Serrata in IBS Subjects With Small Bowel Dysbiosis
Brief Title: Positive Outcomes of the Supplementation With Lecithin-based Delivery Form of Curcuma Longa and of Boswellia Serrata in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0612/22052019
Record Dates: First submitted 2024-04-19; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Boswellia Serrata; Irritable Bowel Syndrome
Keywords: Bloating; Dysbiosis; Boswellia serrata; Curcuma longa; Irritable bowel syndrome; Microbiota; Phytosome
MeSH Terms: conditions — Irritable Bowel Syndrome; Dysbiosis | interventions — turmeric extract; FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CUBO and low FODMAP diet (Intervention) (Active Comparator): Curcuma and Boswellia serrata extract plus a Low Fodmap Diet
  Interventions: Dietary Supplement: Curcuma and boswellia extracts plus low fodmap diet
- LFD (Control) (Other): Only Low Fodmap Diet
  Interventions: Other: Low Foodmap diet

INTERVENTIONS:
Dietary Supplement: Curcuma and boswellia extracts plus low fodmap diet — Low Foodmap diet + Curcuma and boswellia extracts both formulated in sunflower lecithin (Phytosome™) and processed with a strong commitment to sustainability
  Arms: CUBO and low FODMAP diet (Intervention)
Other: Low Foodmap diet — such as lactose or gluten free diet in the last 6 months
  Arms: LFD (Control)

SUMMARY:
Small bowel dysbiosis (SBD), is a frequent finding in subjects with irritable bowel syndrome (IBS). The formula-tion in sunflower lecithin (Phytosome) of Curcuma longa and Boswellia serrata demonstrated beneficial effects on intestinal microbiota. The aim of this study was to evaluate the effect of a lecithin-based delivery formulation of Curcuma longa and of Boswellia serrata extracts (CUBO), on SBD in IBS subjects.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18 to 70 years;
* diagnosis of moderate IBS according to Rome IV criteria;
* dysbiosis of the small bowel, defined by increased urinary indican values with normal values of urinary skatole;
* evidence of abdominal bloating and abdominal pain

Exclusion Criteria:

* normal values of urinary indican or increased values of urinary skatole ;
* subjects who were already on a low FODMAP diet (LFD) or other dietary prescription, such as lactose or gluten free diet in the last 6 months;
* insulin-dependent diabetes or seafood, nuts or soy allergies ;
* positive history of symptomatic diverticular disease, celiac disease, inflammatory bowel disease or microscopic colitis;
* colonic or small bowel or gallbladder surgery ;
* severe vomiting or bloody diarrhea ;
* liver disease (defined as altered values of liver function tests) or severe renal disease (defined as serum creatinine >1.5 mg/dL) or treatment with antibiotics, excluding those for topical use, within the last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of Lecithin formulation on small bowel dysbiosis | from baseline to 30 days
  The primary endpoint was the change of small bowel dysbiosis established by the decrease in urine indican values. The dysbiosis of the small bowel was defined by increased urinary indican values with normal values of urinary skatole.
  Urinary values of indican (3-indoxyl sulfate) were evaluated through a colorimetric method. Urinary indican was considered normal when the levels were lower than 10 mg/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Mariangela Rondanelli, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No